CLINICAL TRIAL: NCT02051465
Title: A Randomized Controlled Trial to Evaluate Effectiveness and Safety of the Endoscopic Removal of Large and Flat Colonic Polyps With LumenR RetractorTM (LR) as a Modified Colonic Overtube
Brief Title: Effectiveness and Safety of the Endoscopic Removal of Large and Flat Colonic Polyps With LumenR RetractorTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Principal Investigator, Sergey Kantsevoy, Director of Therapeutic Endoscopy, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC 2012-64
Record Dates: First submitted 2014-01-26; First posted 2014-01-31 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Colonic Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LumenR Retractor (Experimental): Endoscopic removal of polyp using modified overtube LumenR Retractor
  Interventions: Device: LumenR Retractor
- Removal without overtube (Active Comparator): Endoscopic removal of polyp without overtube
  Interventions: Device: Removal without overtube

INTERVENTIONS:
Device: LumenR Retractor — Polyp removal using LumenR Retractor Modified overtube
  Arms: LumenR Retractor
Device: Removal without overtube — Endoscopic removal of polyp without overtube
  Arms: Removal without overtube

SUMMARY:
Colorectal cancer accounted for 142,570 new cancer cases and 51,370 cancer deaths in USA in 2010 and worldwide has become the third most common cancer and second leading cause of cancer related deaths. Colonic adenomatous polyps are known precursors of colorectal cancer and endoscopic removal of the polyps prevents development of colon cancer.

Removal of such large polyps requires special endoscopic techniques-endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD), which are more technically difficult to perform, labor intensive, time consuming and carries higher risks of complications (bleeding, perforations, etc.). The purpose of this study is to determine the effectiveness and safety of the LumenR Retractor in performing EMR and ESD. It is hypothesized that the use of this modified colonic overtube will simplify colonoscopic removal of difficult polyps, decrease the time needed to complete the procedure and decrease the rate of complications post endoscopic removal of large and flat colonic.

DETAILED DESCRIPTION:
All patients presented for endoscopic removal of difficult colonic polyps will be eligible for the study based on inclusion and exclusion criteria. All procedures will be explained by the Investigator and all subjects undergoing treatment will review and sign the study Informed Consent prior to the procedure. Each subject will be randomly assigned to two groups, Group 1 and Group 2, and according to the assignment, the LumenR Retractor will be used or not during the procedure.

Patient preparation, including intravenous sedation, will be the same for both Groups.

Group 1: A traditional pediatric colonoscope will be advanced into the colon and endoscopic removal of the polyp will be performed.

Group 2: A traditional pediatric colonoscope with a modified overtube preloaded over the endoscope will be advanced into the colon. After the polyp is reached, the overtube will be advanced forward and expanded around the polyp. Endoscopic removal of the polyp with the use of commercially available graspers and biopsy forceps inserted through the overtube working channels will be performed.

At the conclusion of each procedure, the size of the polyp, total procedure time, amount of CO2 used for colonic insufflation, amount of fluid used for submucosal injection, and any complications, including bleeding and perforation, will be recorded. At the end of the procedure, if necessary, the resulting mucosal defect after lesion removal will be closed with endoscopic clips or endoscopic suturing device.

After completion of procedure, all subjects will be recovered according to standard recovery room protocol and then discharged home or admitted to hospital if necessary. Subjects will be followed at 24 hours, and 10 days post treatment and any complications post endoscopic removal of the polyp will be recorded. At 3 months post treatment, all subjects will have repeat colonoscopy to evaluate post polypectomy site and remove any residual polypoid tissue found.

ELIGIBILITY:
Inclusion Criteria:

* Colonic polyps 2cm in size or greater
* Subject 17 to 90 years of age
* Female subjects must have negative pregnancy test within last 24 hours timeline, and no intentions to become pregnant or be sterilized during participation in study.

Exclusion Criteria:

* Colonic polyps less than 2cm in size
* Under 17 or over 90 years of age
* Unwilling to consent or comply with protocol requirements
* Uncorrectable bleeding disorders (INR more than 1.5; platlet count less than 50,000)
* Allergy to materials from which the device is constructed- Polyvinyl Chloride, Nitinol, Watershed, Polycarbonate, and Polytetrafluoroethylene
* Received experimental drug or device within 3 months prior to start of study
* Treatment with an investigational drug or medical device during the study period
* Female subjects that are pregnant or lactating or intending to become pregnant during the period of the study, or who would not use an adequate method of contraception (contraceptive pill, intra-uterine device) for the duration of the study
* Psychological condition, or under treatment for any condition which, in the opinion of the Investigator and/or consulting physician(s), would constitute an unwarranted risk

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of successful en block removal of polyps | 1 year
Length of time required to remove large and flat colonic polyps | Day 1

SECONDARY OUTCOMES:
Amount of carbon dioxide (CO2) gas for colonic insufflation used during procedure | Day 1
Amount of solution used for submucosal injection to lift the polyp | Day 1
Presence of residual polypoid tissue at the site of polypectomy | 3 months
  A colonoscopy will be performed to evaluate the polypectomy site and remove any residual polypoid tissue if found.
Safety assessment based on the number of delayed adverse events and complications | 10 days
Rate of bleeding during polypectomy | 1 year
  Estimate of rate of bleeding during endoscopic removal of difficult colonic polyps
Rate of perforation during polypectomy | 1 year
  To compare rate of perforation during endoscopic removal of difficult colonic polyps

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Kantsevoy, M.D., Ph.D., Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States